CLINICAL TRIAL: NCT04306185
Title: Ovarian Fragmentation Study (Crespo Medical Team)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Equipo Juana Crespo (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fibrotomia1
Record Dates: First submitted 2020-03-06; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Ovarian Failure; Premature Ovarian Failure; IVF
Keywords: ovarian fragmentation; Kawamura; ovarian rejuvenation
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OVARIAN FRAGMENTATION (Experimental): Ovarian fragmentation through laparoscopy in patients who meet criteria ( Poor ovarian responders and poor ovarian reserve).
  Interventions: Procedure: OVARIAN FRAGMENTATION

INTERVENTIONS:
Procedure: OVARIAN FRAGMENTATION — BILATERAL OVARIAN CORTEX FRAGMENTATION USING LAPAROSCOPIC SCISSORS

SUMMARY:
This is a study designed to validate Kawamura´s theory and investigation of activation of primordial follicles through ovarian cortex fragmentation. Our aim is to evaluate embryo quality following this procedure in poor ovarian responders and patients with decreased ovarian reserve. Secondary objectives are to assess potential association with the number of oocytes retrieved and pregnancy rates after IVF.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal surgery need for fertility cause.
* Bad embryo quality (>2 cycles with < 1 embryo A-B quality. With:

A. Poor ovarian responders (previous ≤ 3 retrieved metaphase II oocytes) in a conventional cycle.

B. Decreased ovarian reserve (antral follicle count (AFC) ≤ 5 or antiMullerian hormone (AMH) ≤ 0.5 ng/mL).

C.Premature ovarian insufficiency according to:

* Patients < 40 years old.
* At least 1 year of amenorrhea.
* Follitropin serum levels (FSH) >35 IU/ml in two serum samples separated by at least 1 month.
* Estradiol serum levels (E2) < 20 pg/mL.

Exclusion Criteria:

1. Clinical/ultrasonographical signs of severe endometriosis ( or endometrioma).
2. Age over 45 years (EMC)
3. Previous ovarian/pelvic surgery. Unilateral oophorectomy.
4. Body Mass Index > 30
5. Previous gonadotoxic treatment.
6. Genito-urinary tract malformations.
7. Inform consent unsigned.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Embryo quality improvement following ovarian fragmentation (Using ASEBIR Embryo Classification, 2015) | 1 year
  Embryo quality improvement following ovarian cortex fragmentation in poor ovarian responders or patients with premature ovarian insufficency using ASEBIR Classification (2015).

SECONDARY OUTCOMES:
- Follicle growth rate before and after ovarian cortex fragmentation. | 2 months.
  Number of antral Follicles in IVF treatment before ovarian fragmentation and after IVF following ovarian fragmentation.
- Oocyte number and M-II oocyte (mature oocytes) before and after ovarian cortex fragmentation. | 2 months
- AntiMullerian hormone (AMH) serum levels before and two months after the procedure. | 2 months.
- Number of embryos before and after ovarian cortex fragmentation. | 2 months
- Clinical pregnancy rate following ovarian cortex fragmentation. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ander Morales Vicente, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Revelli A, Marchino G, Dolfin E, Molinari E, Delle Piane L, Salvagno F, Benedetto C. Live birth after orthotopic grafting of autologous cryopreserved ovarian tissue and spontaneous conception in Italy. Fertil Steril. 2013 Jan;99(1):227-230. doi: 10.1016/j.fertnstert.2012.09.029. Epub 2012 Oct 23. PMID 23102860
- [Background] Isachenko V, Isachenko E, Keck G, Dittrich R, Montag M, van der Ven H, Mallmann P, Muller A, Distler W, Beckmann MW, Rahimi G. First live birth in germany after re-transplantation of cryopreserved ovarian tissue: original device for initiation of ice formation. Clin Lab. 2012;58(9-10):933-8. PMID 23163109
- [Background] Baird DT, Webb R, Campbell BK, Harkness LM, Gosden RG. Long-term ovarian function in sheep after ovariectomy and transplantation of autografts stored at -196 C. Endocrinology. 1999 Jan;140(1):462-71. doi: 10.1210/endo.140.1.6453. PMID 9886858
- [Background] Donnez J, Dolmans MM, Demylle D, Jadoul P, Pirard C, Squifflet J, Martinez-Madrid B, Van Langendonckt A. Restoration of ovarian function after orthotopic (intraovarian and periovarian) transplantation of cryopreserved ovarian tissue in a woman treated by bone marrow transplantation for sickle cell anaemia: case report. Hum Reprod. 2006 Jan;21(1):183-8. doi: 10.1093/humrep/dei268. Epub 2005 Aug 25. PMID 16126712
- [Background] Callejo J, Salvador C, Gonzalez-Nunez S, Almeida L, Rodriguez L, Marques L, Valls A, Lailla JM. Live birth in a woman without ovaries after autograft of frozen-thawed ovarian tissue combined with growth factors. J Ovarian Res. 2013 May 7;6(1):33. doi: 10.1186/1757-2215-6-33. PMID 23647552
- [Background] Kawamura K, Kawamura N, Hsueh AJ. Activation of dormant follicles: a new treatment for premature ovarian failure? Curr Opin Obstet Gynecol. 2016 Jun;28(3):217-22. doi: 10.1097/GCO.0000000000000268. PMID 27022685
- [Result] Donnez J, Jadoul P, Pirard C, Hutchings G, Demylle D, Squifflet J, Smitz J, Dolmans MM. Live birth after transplantation of frozen-thawed ovarian tissue after bilateral oophorectomy for benign disease. Fertil Steril. 2012 Sep;98(3):720-5. doi: 10.1016/j.fertnstert.2012.05.017. Epub 2012 Jun 13. PMID 22698640